CLINICAL TRIAL: NCT06581614
Title: Effect of Implant Supported Fixed Restoration on Masticatory Efficiency in Patients With Second Molar Loss
Brief Title: Masticatory Performance Evaluation
Acronym: MPE
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202407119RINA
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Masticatory Performance
Keywords: implant supported fixed prosthesis; masticatory efficiency; chewing gum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective group: Patients who have lost their second molar, are scheduled to undergo single-implant reconstruction at the Prosthodontics Department of National Taiwan University Hospital, and do not have any major physical or mental health conditions
  Interventions: Diagnostic Test: masticatory function test
- retrospective group: Patients who have lost their second molar, have undergone single-implant-supported fixed restoration reconstruction at the Prosthodontics Department of National Taiwan University Hospital, and do not have any major physical or mental health conditions.
  Interventions: Diagnostic Test: masticatory function test

INTERVENTIONS:
Diagnostic Test: masticatory function test — During the test, participants will be given a piece of chewing gum to assess their masticatory function when the second molar implant-supported fixed denture is in place.

SUMMARY:
The purpose of this experiment is to combine research on masticatory efficiency with the reconstructive expertise of the prosthodontics clinic, focusing on implant-supported fixed dentures as the contemporary gold standard for reconstruction. The goal is to investigate the impact of such prosthetic reconstructions on masticatory efficiency. We will invite patients who have lost their second molar and have undergone single-implant-supported fixed denture reconstruction at the Prosthodontics Department of National Taiwan University Hospital to participate in masticatory function tests. The tests will use a new and relatively simple chewing gum, with the aim of enhancing patients' masticatory function through implant reconstruction in a clinical setting, thereby improving patient well-being and understanding of dental implants. On the research side, the study aims to provide guidance for strategies in the reconstruction of masticatory function.

DETAILED DESCRIPTION:
Chewing is one of the important steps in the process of food digestion, and it is crucial for human nutritional intake and oral health. Chewing efficiency relates to the ability to eat and is influenced by many factors, with the key factor being the absence of posterior teeth. According to traditional occlusal theory, the anterior teeth guide and act as a facade, while the posterior teeth provide support and chewing function. The loss of posterior teeth leads to a decrease in chewing efficiency. In 1954, Dr. A. Albert Yurkstas and others proposed that in healthy adults, the loss of the first molar results in a 33% decrease in chewing efficiency; the loss of the second and third molars results in a 44% decrease; and the loss of the first, second, and third molars results in a 78% decrease. This study laid the foundation for understanding how tooth loss leads to decreased chewing efficiency and highlights the goal of prosthodontics to restore dental arches and chewing function to benefit people.

The purpose of this experiment is to combine the study of chewing efficiency with the expertise of prosthodontics in reconstruction, aiming to investigate the impact of contemporary gold-standard artificial implant-supported fixed restorations on chewing efficiency. The study invites patients missing the second molar and those receiving implant-supported fixed prostheses reconstruction in the Department of Prosthodontics at National Taiwan University Hospital. The new and simpler color-changeable chewing gum will be used to test their chewing efficiency. This will explore the importance of implant-supported fixed prostheses in reconstructing chewing function after the loss of the second molar, aiming to improve patient well-being and understanding of dental implants by restoring chewing function through clinical implant reconstruction. In the research field, this study provides guidance for the reconstruction strategies of chewing function

ELIGIBILITY:
For prospective group:

Inclusion Criteria:

* Patients who have lost their second molar, are scheduled to undergo single-implant reconstruction at the Prosthodontics Department of National Taiwan University Hospital, and do not have any major physical or mental health conditions.

Exclusion Criteria:

* Severe temporomandibular joint disorder
* Inability to comply with the treatment schedule
* Inability to cooperate with masticatory function tests
* Lack of opposing teeth for the implant-supported restoration
* Patients whose anterior teeth will be included in the prosthetic reconstruction or whose occlusion will undergo significant changes after reconstruction

For retrospective group:

Inclusion Criteria:

* Patients who have lost their second molar, have undergone single-implant-supported fixed restoration reconstruction at the Prosthodontics Department of National Taiwan University Hospital, and do not have any major physical or mental health conditions.

Exclusion Criteria:

* Implant-supported dentures that cannot be removed or have significant damage
* Severe temporomandibular joint disorder
* Inability to comply with the treatment schedule
* Inability to cooperate with masticatory function tests
* Lack of opposing teeth for the implant-supported denture

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have lost their second molar
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
the masticatory performance of patients | After second molar implant reconstruction was done(at least 1 month after reconstruction)
  During the test, participants will be given a piece of chewing gum to assess their masticatory function when the second molar implant-supported fixed restoration is in place.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hao Lan, Study Director — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Yi-Hao Lan, Taipei

IPD SHARING:
Plan to Share IPD: No
For the privacy of patients

REFERENCES:
- [Result] Tarkowska A, Katzer L, Ahlers MO. Assessment of masticatory performance by means of a color-changeable chewing gum. J Prosthodont Res. 2017 Jan;61(1):9-19. doi: 10.1016/j.jpor.2016.04.004. Epub 2016 May 17. PMID 27211494